CLINICAL TRIAL: NCT03953417
Title: Pilot Accelerated Theta Burst Stimulation in Treatment-Resistant Bipolar Depression
Brief Title: Pilot Accelerated Theta Burst in Treatment-Resistant Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ian Kratter, Clinical Assistant Professor, Department of Psychiatry and Behavioral Sciences, Stanford University Medical Center, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49486
Record Dates: First submitted 2019-04-18; First posted 2019-05-16 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression
Keywords: Bipolar Disorder; Treatment Resistant Depression; Transcranial Magnetic Stimulation (TMS); Theta Burst
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated intermittent theta burst treatment (Experimental): All participants will receive accelerated intermittent theta-burst stimulation.
  Interventions: Device: Accelerated intermittent theta-burst treatment

INTERVENTIONS:
Device: Accelerated intermittent theta-burst treatment — All participants will receive accelerated intermittent theta-burst stimulation to the left DLPFC. Treatment will be targeted by utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of resting motor threshold adjust to the skull to cortical surface distance.
  Stimulation will be delivered to left DLPFC using the MagPRo stimulator.

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for treatment-resistant bipolar depression. In this open-label study, all participants will receive accelerated theta-burst stimulation.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 minutes over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been very successful in real-world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session over 4-6 weeks). Recently, researchers have aggressively pursued modifying the treatment parameters to reduce treatment times with some preliminary success. In a recent study, the investigators applied this accelerated paradigm in individuals with treatment-resistant depression (TRD), which showed a significant antidepressant effect (90% remission rate). Additionally, 3 participants from this study carried a bipolar TRD diagnosis and responded at minimum, equally as well, with no adverse events experienced or manic/hypomanic conversion observed during the treatment series. This study intends to further modify the parameters to create a more rapid form of this treatment for bipolar TRD, and look at the change in clinical measures and neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 80 years of age.
* Able to provide informed consent.
* Diagnosed with Bipolar Disorder and currently experiencing a Major Depressive Episode (MDE).
* Meet the threshold on the total MADRS score of >/=20 at baseline.
* In good general health, as ascertained by medical history.
* If female, a status of non-childbearing potential or use of an acceptable form of birth control.
* History of rTMS failure with FDA approved rTMS parameters is permitted.

Exclusion Criteria:

* Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
* Female that is pregnant or breastfeeding.
* Female with a positive pregnancy test at participation.
* Total MADRS score of < 20 at study entry.
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR), with the exception of nicotine dependence.
* Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).
* History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their bipolar depression or has been predominant to their bipolar depression at any time within six months prior to screening.
* Considered at significant risk for suicide during the course of the study.
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
* History of positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.
* Current (or chronic) use of opiates.
* History of epilepsy.
* History of shrapnel or metal in the head or skull.
* History of cardiovascular disease or cardiac event.
* History of OCD.
* History of autism spectrum disorder.
* Current psychosis
* Any change in medication of which the study PI is not aware of.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Kratter, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
clintrials.gov

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Fox MD, Snyder AZ, Vincent JL, Corbetta M, Van Essen DC, Raichle ME. The human brain is intrinsically organized into dynamic, anticorrelated functional networks. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9673-8. doi: 10.1073/pnas.0504136102. Epub 2005 Jun 23. PMID 15976020
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396

RESULTS

PARTICIPANT FLOW:
Groups:
- Accelerated Intermittent Theta Burst Treatment: All participants will receive accelerated intermittent theta-burst stimulation.
  Accelerated intermittent theta-burst treatment: All participants will receive accelerated intermittent theta-burst stimulation to the left DLPFC. Treatment will be targeted by utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of resting motor threshold adjust to the skull to cortical surface distance.
  Stimulation will be delivered to left DLPFC using the MagPRo stimulator.
Period: Overall Study
Arm/Group | Accelerated Intermittent Theta Burst Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Accelerated Intermittent Theta Burst Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 41 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Montgomery Asberg Depression Rating Scale (MADRS)
Description: A ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  The MADRS consists of ten questions. Each interview question is rated from 0 to 6 with an overall score of 60 or less. Higher scores indicate increasing depressive symptoms. A total score of 0 to 6 indicates the absents of depressive symptoms, 7 to 19 indicates mild depressive symptoms, 30 to 34 indicates moderate depressive symptoms, 35 to 60 indicates severe depressive symptoms.
Time Frame: Baseline and immediately post-treatment (6 days post baseline)
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accelerated Intermittent Theta Burst Treatment
Number analyzed (Participants) | 7
score on a scale
  Baseline | 40.0 (9.8)
  Immediate Post Treatment: number analyzed (Participants) | 6
  Immediate Post Treatment | 5.7 (10.7)

2. Secondary Outcome: Change From Baseline Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition.
  There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. The overall total score is a maximum of 60.
  Typical YMRS baseline scores can vary a lot. They depend on the patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2).
Time Frame: Baseline and immediate post-treatment (6 days post baseline)
Population: Participants with data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accelerated Intermittent Theta Burst Treatment
Number analyzed (Participants) | 5
score on a scale
  Baseline | 0.8 (1.8)
  Immediate Post Treatment: number analyzed (Participants) | 4
  Immediate Post Treatment | 0 (0)

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Accelerated Intermittent Theta Burst Treatment
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
There are no limitations and caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03953417/Prot_000.pdf